CLINICAL TRIAL: NCT01241539
Title: Open Label, Non Randomized, Multiple Dose Phase I Study to Investigate the Elimination, Pharmacokinetics, Pharmacodynamics and Safety of Dabigatran Etexilate (Pradaxa) Under Steady State Conditions Before, During and After Haemodialysis in Patients With End Stage Renal Disease (ESRD) Undergoing Regular Haemodialysis
Brief Title: Pharmacokinetics of Dabigatran Etexilate (Pradaxa®) During Haemodialysis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 1160.121; 2010-021819-16 (EudraCT Number: EudraCT)
Record Dates: First submitted 2010-11-15; First posted 2010-11-16 (Estimated); Results first posted 2012-07-27 (Estimated); Last update posted 2014-04-07 (Estimated); Status verified 2014-02

CONDITIONS: Cardiovascular Diseases; Kidney Failure, Chronic
MeSH Terms: conditions — Cardiovascular Diseases; Kidney Failure, Chronic | interventions — Dabigatran

ARMS (3):
- Dabigatran etexilate 110 mg (Experimental): Capsule, oral
  Interventions: Drug: Dabigatran etexilate
- Dabigatran etexilate 75 mg (Experimental): Capsule, oral
  Interventions: Drug: Dabigatran etexilate
- Dabigatran etexilate 150 mg (Experimental): Capsule, oral
  Interventions: Drug: Dabigatran etexilate

INTERVENTIONS:
Drug: Dabigatran etexilate — 150 mg capsule
  Arms: Dabigatran etexilate 150 mg
Drug: Dabigatran etexilate — 75 mg capsule
  Arms: Dabigatran etexilate 75 mg
Drug: Dabigatran etexilate — 110 mg capsule
  Arms: Dabigatran etexilate 110 mg

SUMMARY:
The current study will allow the assessment of pharmacokinetics, pharmacodynamics, elimination rate and clearance of dabigatran etexilate during and following haemodialysis in ESRD patients.

ELIGIBILITY:
Inclusion criteria:

* End stage renally disease (ESRD), undergoing haemodialysis
* ESRD patients in relatively good health
* Age 21 - 60 years inclusive
* Signed and dated written informed consent prior to admission to the study

Exclusion criteria:

* Clinically relevant laboratory or physical examination abnormalities (except for renal function tests or deviation of clinical laboratory values) that are related to renal impairment
* Moderate and severe concurrent liver function impairment
* Surgery of gastrointestinal tract (except appendectomy or herniotomy) or evidence of significant gastrointestinal motility problems
* Recent or contemplated diagnostic or therapeutic procedures with potential for uncontrollable bleeding
* Intake of medication, which influences the blood clotting
* Subjects not able to understand and comply with protocol requirements, instructions and protocol-stated restrictions
* For women with childbearing potential: no reliable contraception
* Participation in another trial with an investigational drug (<2 months prior to administration or during trial)
* Scheduled to receive a donor kidney transplant during the course of the study

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2010-11; Primary Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1160.121.1 Boehringer Ingelheim Investigational Site, Berlin, Germany

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was an open-label, 2-period, fixed-sequence, multiple dose trial. On Day 1, all patients were treated with Dabigatran 150 mg, on day 2, with 110 mg at 10:00, and on day 3, 75 mg 8 h before dialysis. The target blood flow rate on day 3 of period 1 was 200mL/min, whilst that in period 2 was 400mL/min.
Groups:
- Dabigatran: Period 1 target blood flow rate during dialysis was 200mL/min. Period 2 target blood flow rate during dialysis was 400mL/min.
Period: Period 1
Arm/Group | Dabigatran
Started | 7
Completed | 7
Not Completed | 0
Period: Period 2
Arm/Group | Dabigatran
Started | 7 (After a wash-out phase of at least 6 weeks.)
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS) included all 7 subjects who were dispensed trial medication and were documented to have taken at least 1 dose of investigational treatment.
Groups:
- Dabigatran: Dabigatran treated patients
Arm/Group | Dabigatran
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.3 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 7

OUTCOME MEASURES:

1. Primary Outcome: Dialysis Clearance of Dabigatran
Description: Dialysis clearance of dabigatran from blood (CLD,b) and dialysis clearance of dabigatran from plasma (CLD) were calculated and indicate how quickly dabigatran is cleared out from blood or plasma.
Time Frame: 4 hours
Population: Pharmacokinetic set (PKS) includes all evaluable patients of the treated set who received at least one dose of dabigatran etexilate and who provide at least one observation for at least one Pharmacokinetic (PK) endpoint without important protocol violations relevant to the evaluation of PK.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Groups:
- Dabigatran P1: Period 1 target blood flow rate during dialysis was 200mL/min
- Dabigatran P2: Period 2 target blood flow rate during dialysis was 400mL/min
Arm/Group | Dabigatran P1 | Dabigatran P2
Number analyzed (Participants) | 7 | 7
mL/min
  Total dabigatran clearance (CLD,b) from blood | 161 (5.01) | 241 (3.08)
  Total dabigatran clearance (CLD) from plasma | 120 (5.09) | 183 (4.30)
  Free dabigatran clearance (CLD,b) from blood | 167 (4.60) | 251 (2.17)
  Free dabigatran clearance (CLD) from plasma | 124 (4.48) | 190 (3.68)

2. Primary Outcome: Extent Cleared From Circulation (Plasma) During 1 Complete Cycle of Dialysis
Description: Extent of dabigatran that is removed from blood during one complete 4-hour cycle of dialysis was computed by the difference of plasma concentration at the start and at the end of dialysis relative to the start concentration and is therefore measured as a percentage.
Time Frame: 4 hours
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage
Arm/Group | Dabigatran P1 | Dabigatran P2
Number analyzed (Participants) | 7 | 7
Percentage
  Total Dabigatran | 48.8 (10.9) | 59.3 (6.69)
  Free Dabigatran | 49.7 (9.10) | 59.3 (6.13)

3. Primary Outcome: Plasma Concentration Extraction Ratio
Description: Plasma concentration extraction ratio was measured directly at the dialysis machine and computed as the difference of the predialysis plasma concentration and the postdialysis plasma concentration relative to the predialysis concentration on the percentage scale (minimum: 0 percent of extraction (worst), maximum: 100 percent of extraction).
Time Frame: 4 hours
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage
Arm/Group | Dabigatran P1 | Dabigatran P2
Number analyzed (Participants) | 7 | 7
Percentage
  Total Dabigatran | 79.9 (9.01) | 61.4 (9.54)
  Free Dabigatran | 82.6 (8.21) | 63.7 (8.60)

4. Secondary Outcome: Area Under the Curve Exposure to Dabigatran During the First 8 Hours Post Dose (AUC0-8h)
Description: Area under the concentration-time curve of total and free dabigatran in plasma over the time interval from 0 to 8 hours after the second and third administration of dabigatran.
Time Frame: Days 2 and 3
Population: Pharmacokinetic set (PKS) includes all evaluable patients of the TS who received at least 1 dose of dabigatran etexilate, who provided at least 1 observation for at least 1 Pharmacokinetics (PK) endpoint, and who did not have important protocol violations relevant to the evaluation of PK
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Dabigatran P1 | Dabigatran P2
Number analyzed (Participants) | 7 | 7
ng*hr/mL
  Total Dabigatran on Day 2 | 1230 (57.1) | 1140 (39.4)
  Total Dabigatran on Day 3 | 1280 (54.4) | 1180 (50.2)
  Free Dabigatran on Day 2 | 907 (51.6) | 802 (44.1)
  Free Dabigatran on Day 3 | 839 (41.3) | 752 (58.0)

5. Secondary Outcome: Maximum Plasma Concentrations of Dabigatran (Cmax)
Description: Maximum measured concentration of total and free dabigatran in plasma after the second and third administration of dabigatran.
Time Frame: Days 2 and 3
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Dabigatran P1 | Dabigatran P2
Number analyzed (Participants) | 7 | 7
ng/mL
  Total Dabigatran on Day 2 | 194 (53.1) | 171 (36.2)
  Total Dabigatran on Day 3 | 176 (54.1) | 159 (50.2)
  Free Dabigatran on Day 2 | 150 (47.3) | 126 (38.1)
  Free Dabigatran on Day 3 | 119 (43.7) | 105 (57.3)

6. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax)
Description: Time to maximum plasma concentration of total and free dabigatran in plasma after the third administration of dabigatran.
Time Frame: Day 3
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | Dabigatran P1 | Dabigatran P2
Number analyzed (Participants) | 7 | 7
h
  Total Dabigatran | 1.49 (38.4) | 2.13 (74.1)
  Free Dabigatran | 1.35 (38.4) | 1.83 (27.3)

7. Secondary Outcome: Coagulation Parameters
Description: Assessment of blood coagulation parameters 'activated partial thromboplastin time' (aPTT) and 'factor IIa inhibition' (anti-FIIa) measured with the diluted thrombin time assay. Time to the formation of a fibrin clot (coagulation) is measured in seconds.
Time Frame: Day 3
Population: TS
Measure: Mean (Standard Deviation); unit: sec
Arm/Group | Dabigatran P1 | Dabigatran P2
Number analyzed (Participants) | 7 | 7
sec
  Activated partial thromboplastin time (aPTT) | 46.91 (12.22) | 44.26 (10.98)
  Factor IIa inhibition (anti-FIIa) | 43.27 (7.99) | 43.09 (5.38)

8. Secondary Outcome: Safety and Tolerability
Description: Tolerability refers to the number of non-tolerable patients as assessed through the subjective examination of adverse events (AE). Safety refers to the number of patients with treatment emergent AEs. These numbers are presented on the overall Dabigatran treatment.
Time Frame: 2 periods of 5 days each
Population: TS
Measure: Number; unit: Participants
Arm/Group | Dabigatran
Number analyzed (Participants) | 7
Participants
  Treatment emergent adverse events | 2
  Assessment of tolerability by the investigator | 0

9. Secondary Outcome: Additional Safety Parameters
Description: By study design abnormalities could be due to dialysis or Dabigatran.
Time Frame: 2 periods of 5 days each
Population: TS
Measure: Number; unit: Participants
Arm/Group | Dabigatran
Number analyzed (Participants) | 7
Participants
  Electrocardiogram (ECG) abnormalities | 0
  Vital sign abnormalities | 0
  Physical finding abnormalities | 0
  Laboratory abnormalities: Haematology | 0
  Laboratory abnormalities: Clinical chemistry | 0

ADVERSE EVENTS:
Time Frame: 2 periods of 5 days each
Description: Before and after dialysis
Arm/Group | Dabigatran
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 2/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dabigatran (N=7)
Headache (Nervous system disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.